CLINICAL TRIAL: NCT06501300
Title: Tuning in to Kids in School - Competence Building and Collaboration in the Team Around Primary School Students
Acronym: TIKiS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sophie Havighurst (Other)
Collaborators: University of Melbourne (Other); University of Stavanger (Other)
Responsible Party: Sponsor-Investigator, Sophie Havighurst, Principal Investigator, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: TIKiS Norway
Record Dates: First submitted 2024-02-05; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Teachers; Schools; Tuning in to Kids; Intervention; TIK; TIKiS; Emotion Socialisation; Emotional Competence
MeSH Terms: interventions — Schools

STUDY DESIGN:
Intervention Model Description: 10 schools are assigned to a wait-list control group, while 10 are assigned to the intervention group.
Who Masked: Outcomes Assessor
Masking Description: Observers do not know whether the schools they visit are intervention or control schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Teachers and relevant school staff six 90-minute supervised group lessons with a 1-2 week space between each time.
  School leaders attend three 90-minute sessions adapted to them
  Interventions: Behavioral: Emotion-focused: Tuning in to Kids in School
- Waitlist Control (No Intervention): Receives no intervention, business as usual. Receives intervention the following year.

INTERVENTIONS:
Behavioral: Emotion-focused: Tuning in to Kids in School — The aim of the TIKiS is to improve emotion coaching and reduce emotion dismissing in elementary school teachers through six x 90-minute group sessions.
  Arms: Intervention

SUMMARY:
The current project is a randomized controlled trial of the Australian evidence-based parenting program Tuning in to Kids® which has been adapted for using with Norwegian elementary school teachers (Tuning in to Kids in Schools; TIKiS).

TIKiS aims to improve emotion socialization practices of primary school teachers so that children's emotional competence is promoted.

This project will determine effectiveness and implementation quality of TIKiS through questionnaire and observation measures given before and after the intervention, comparing intervention and wait-list control schools.

DETAILED DESCRIPTION:
This project is a collaboration between the University of Oslo, the education agency and health agency in Oslo municipality, Norway.

A total of 20 schools will be recruited for the project, and randomly allocated to the intervention or wait-list control condition (10 in each). Teachers in the intervention schools will receive the TIKiS intervention delivered by trained facilitators. Facilitators of the teacher groups will be from staff from education and health agencies and will have at least a masters' degree in psychology, pedagogy or similar.

The TIKiS program facilitators attend a two day training in TIKiS. In addition, they will attend a 90-minute workshop and receive three days of 90-minute program supervision before they act as program facilitators for the teachers.

In the intervention condition, school leaders will attend adapted three 90-minute group sessions to assist with implementation. All teachers in the intervention schools will attend introduction sessions outlining the program. Then teachers and other relevant school staff (special education teachers, resource teachers, social teachers and assistants) in grade 1-4 (the first 4 years of elementary school) will attend six x 90 minute group sessions led by a pair of program facilitators.

In intervention and control schools, facilitators of groups, teachers and relevant school staff will complete questionnaires at baseline and follow-up. Observations of classes of these teachers and staff will be conducted at baseline and follow-up.

Control schools will receive the intervention following completion of all follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* School staff that work with children in grades 1.-4.

Exclusion Criteria:

* (Exclusion from analysis) school staff in the intervention school that did not participate in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Classroom Assessment Scoring system - CLASS- K3 | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A structured, validated observation measure of a classroom's social-emotional environment. Scored from 1 to 7 where 1 is low score (few behaviour markers observed or are rarely observed) and 7 is a high score (many behaviour indicators are frequently observed). (Pianta, La Paro, & Hamre, 2008).
Coping with Children's Negative Emotions Teacher Version - CCNES-T: | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A measure of emotion coaching and emotion dismissing behaviors (Fabes et al., 2000). This study uses a short form of the original CCNES (21 questions), which has been modified and translated to Norwegian.
  Teachers rate how likely they are to respond to childrens' expressions of negative emotions in various scenarios on a scale of 1 (very unlikely) to 7 (very likely).
Program differentiation | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  Program differentiation is how differnt our intervention is from similar interventions that the school has used recently. This is measured by asing teachers to what degree they have worked with similar teaching strategies in the previous year on a scale of 1 (not at all) to 5 (a lot).
Content Fidelity/Adherance | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  Content Fidelity/Adherance is is how much of the manual and planned content that the facilitators cover for each group session. Facilitators fill in a checklist of core components after each group session to get the proportion of core content completed for each session and in total for the whole intervention.
Dosage | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  Dosage is how much of the intervention each participant received, which will be measured as the proportion of intervention sessions that each teacher participated in.
Reach | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  Reach is measured as the proportion of eligible teachers that have participated in the intervention, and the proportion of eligible schools that have participated.
Teacher Implementation | 5 months after intervention (post-intervention)
  Teacher feedback on program satisfaction and use of program content will be measured quantitively trhough a questionnaire and qualitatively and through focus group interviews.
  The questionnaire will ask about obstacles and ease of attending the intervention and using the learned content afterwards, and what aspects they found useful on a scale of 1 to 7 where 1 is a low score and 7 is a high score. The questionnaire will also ask about what cocepts they have used, and what stopped them from attending using multiple choice with a free text option.
  The focus group interviews will be used to get a more detailed assessment of program satisfaction and use of program content

SECONDARY OUTCOMES:
Affect Integration Inventory (AII) | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A measure of how well various emotions are integrated (Solbakken & Monsen, 2017). Teachers rate how well 18 statements about emotions describe them from a scale of 0 (doesnt fit at all) to 9 (fits perfectly).
Bergen burnout inventory (BBI) | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A measure of employee burnout with 9 items. Participants rate how nmuch they agree with each of the 9 statemetns from 1 (disagree completely ) to 6 (agree completely).
  (Matthiesen, 1992; Salmela-Aro et al., 2011)
Hopkins symptom checklist 10 - HSCL-10 | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A measure of distress, which consists of two subscales; anxiety and depression (Derogatis et al., 1974; Hesbacher et al., 1980; Strand et al., 2003). This is a short form of the HSCL with only 10 questions (6 depression, 4 anxiety). Particiapnts rate how much they have experienced each of the 10 symptoms in the past week form 1 (not at all) to 4 (a lot).
Satisfaction with Life scale (SWLS) | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  A 5 item scale that measures satisfaction with life (Diener et al., 1985). Participatns rate how much they agree with each of the 5 statements on a scale of 1 (fits poorly) to 7 (fits perfectly).
Collaboration between school health service, educational psychological services and teachers in Oslo. | Right before intervention (Baseline) and 5 months after intervention (post-intervention)
  Likert scale from 1 to 5 of how well the employees experience the collaboration with the other services. Where 1 is they disagree completely that there is a good collaboration and 5 is they agree completely that there is a good colaboration.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Havighurst, Principal Investigator — University of Oslo
Locations (1):
- Department of Psychology, University of Oslo, Oslo, Norway